CLINICAL TRIAL: NCT02822209
Title: Evaluation of the Impact of a Coordinating Nurse in a Personalized Care Program on Quality of Care, Coordination of the Actors and on Quality of Life for Patients With Lung Cancer. A French Randomized Monocentric Prospective Study
Brief Title: Evaluation of the Impact of a Coordinating Nurse in a Personalized Care Program on Quality of Care, Coordination of the Actors and on Quality of Life for Patients With Lung Cancer
Acronym: EVIDEC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Groupe Hospitalier de la Region de Mulhouse et Sud Alsace (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 804; 2015-A01660-49 (Other: France: Agence Nationale de Sécurité du Médicament et des produits de santé)
Record Dates: First submitted 2016-06-24; First posted 2016-07-04 (Estimated); Last update posted 2019-08-21 (Actual); Status verified 2018-05

CONDITIONS: Lung Cancer
Keywords: coordinating nurse of thoracic oncology; quality of care in thoracic oncology; lung cancer quality of life
MeSH Terms: conditions — Lung Neoplasms | interventions — Nurses, Community Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coordinating nurse added to the personalized care program (Experimental): The coordinating nurse (CN) is dedicated to the newly diagnosed patient to optimize their personalized care program.
  * The CN is the connection between the medical team and the patient. They act according to the instructions from the multidisciplinary staff in charge of bronchopulmonary cancer patients.:
    e.g. Schedule an exam or an hospitalization, collect and share results of useful information to correct treatment's side effects etc
  * Main contact of the patient, the general practitioner and the patient's relatives, they give practical information for the patient's case
  * Quality of life questionnaires - EORTC QLQ-C30 and EORTC QLQ-LC13 - completed by the patient throughout the study.
  * 2 Satisfaction questionnaires completed :
  * satisfaction questionnaire - patient,
  * satisfaction questionnaire - general practitioner or home nurse
  Interventions: Behavioral: EORTC QLQ-C30; Behavioral: Satisfaction questionnaire - patient; Behavioral: Satisfaction questionnaire - general practitioner or home nurse; Behavioral: EORTC QLQ-LC13
- Personalized care program as routine practice (Active Comparator): A personalized care program is decided for the newly diagnosed patient by the multidisciplinary team in charge of lung cancer.
  The care provided will be organized by the medical team, and besides the oncologist, no principal coordinating contact will be in charge of the patient.
  The quality of life questionnaire - EORTC QLQ-C30 and QLQ-LC13 - will be completed by the patient throughout the study.
  * 2 Satisfaction questionnaires completed :
  * satisfaction questionnaire - patient,
  * satisfaction questionnaire - general practitioner or home nurse
  Interventions: Behavioral: EORTC QLQ-C30; Behavioral: Satisfaction questionnaire - patient; Behavioral: Satisfaction questionnaire - general practitioner or home nurse; Behavioral: EORTC QLQ-LC13

INTERVENTIONS:
Behavioral: EORTC QLQ-C30 — Questionnaire submitted at the beginning of the study. Then three more times : 3, 6 and 12 months after the start of anti-cancer therapy. The questionnaire can also be completed before the 12th month: when the care program is about to end
  Other Names: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire
Behavioral: Satisfaction questionnaire - patient — The patient will fill in a satisfaction questionnaire three times : around the third, the sixth and the twelfth month after they started an anti-cancer therapy.
Behavioral: Satisfaction questionnaire - general practitioner or home nurse — The general practitioner or the nurse in charge of the patient at home will fill in a satisfaction questionnaire six months after the patient started an anti-cancer therapy.
Behavioral: EORTC QLQ-LC13 — Questionnaire submitted at the beginning of the study. Then three more times : 3, 6 and 12 months after the start of anti-cancer therapy. The questionnaire can also be completed before the 12th month: when the care program is about to end
  Other Names: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire - Lung Cancer

SUMMARY:
The prognosis of patients with lung cancer is related to the stage of the diagnosis : 73% of one-year-survival rate at stage IA and only 13% one-year-survival rate at stage IV. Controlling the timelines in a care program seems crucial to improve prognosis of lung cancer.

The project aims to evaluate the impact of a coordinating nurse (CN) in a personalized care program for patients of thoracic oncology.

DETAILED DESCRIPTION:
New strategies therapeutics result in a longer survival rate. However their side effects affect the patient's quality of life. Even if these side effects are ambulatory manageable, they require to be treated promptly and tends to increase the active list of patients of the thoracic oncology.

Due to the alteration in the care provided to lung cancer patient, there is a need to coordinate the available means, inside and outside the hospital, to improve the quality of care and the quality of life of the patient.

Every patient of the thoracic oncology department receives a personalized care program as a routine practice. In this study, a coordinating nurse (CN) will be added to the personalized care program. Patients newly diagnosed with a lung cancer will be randomized either in the group with a CN or in the group without a CN.

The study will last one year maximum for each participant. Their quality of life, their satisfaction of the quality of the personalized care program - and their general practitioner's satisfaction - will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient of the thoracic oncology ward between April and November 2016
* Newly diagnosed lung cancer
* Treated in the pneumology ward of the Mulhouse Hospital (France)
* Patient enrolled in another clinical trial can also be enrolled in this study
* Patients who have not disagreed to participate to the study

Exclusion Criteria:

* Secondary cancer in lung
* Relapse of primary cancer in lung of the same histological type
* Previous enrollment in this study
* Uncontrolled psychological problem

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2016-05-11 (Actual); Primary Completion 2017-12-08 (Actual); Study Completion 2017-12-08 (Actual)

PRIMARY OUTCOMES:
Impact of the coordinating nurse on quality of care measured by the variation of timelines in personalized care | At visit 1, around 1 month after the beginning of the study
  Variation of the time between the first appointment with the thoracic oncologist and the first day of anticancer therapy

SECONDARY OUTCOMES:
Analysis of the feedback from healthcare professionals outside the thoracic oncology ward | 6 months after the beginning of the study
  Measured by satisfaction questionnaires submitted to general practitioner or home nurse
Impact of a coordinating nurse in a personalized care program on the patient's quality of life | At the beginning of the study, then around 3, around 6 and around 12 months later
  Evolution of the scoring results of the EORTC QLQ-C30
Impact of a coordinating nurse in a personalized care program on the patient's quality of life | At study enrollment, then around 3 and around 6 and around 12 months later
  Evolution of the scoring results of the EORTC QLQ-LC13
Analysis of the feedback from the patient | Around 3 and around 6 and around 12 months after beginning of study
  Measured by satisfaction questionnaires submitted to the patient

CONTACTS AND LOCATIONS:
Locations (1):
- GHRMSA, Mulhouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martin F, Piquet J, Orlando JP, Blanchon F, Lebas FX. [Clinical research in pneumology in French general hospitals]. Rev Mal Respir. 2014 Nov;31(9):801-3. doi: 10.1016/j.rmr.2014.10.726. Epub 2014 Nov 5. No abstract available. French. PMID 25433584
- [Background] Locher C, Debieuvre D, Coetmeur D, Goupil F, Molinier O, Collon T, Dayen C, Le Treut J, Asselain B, Martin F, Blanchon F, Grivaux M. Major changes in lung cancer over the last ten years in France: the KBP-CPHG studies. Lung Cancer. 2013 Jul;81(1):32-8. doi: 10.1016/j.lungcan.2013.03.001. Epub 2013 Mar 29. PMID 23541463
- [Background] Grivaux M, Locher C, Bombaron P, Collon T, Coetmeur D, Dayen C, Debieuvre D, Goupil F, Le Treut J, Martin F, Molinier O, Asselain B, Zureik M, Blanchon F. [Study KBP-2010-CPHG: inclusion of new cases of primary lung cancer diagnosed in general hospital pneumology departments between 1st January and 31 December 2010]. Rev Pneumol Clin. 2010 Dec;66(6):375-82. doi: 10.1016/j.pneumo.2010.08.001. Epub 2010 Dec 3. French. PMID 21167448
- [Background] Leveque N, Brouchet L, Lepage B, Hermant C, Bigay-Game L, Plat G, Dahan M, Riviere D, Didier A, Mazieres J. [An analysis of treatment delays of thoracic cancers: a prospective study]. Rev Mal Respir. 2014 Mar;31(3):208-13. doi: 10.1016/j.rmr.2013.10.001. Epub 2013 Oct 28. French. PMID 24680111
- [Background] Goldstraw P, Crowley J, Chansky K, Giroux DJ, Groome PA, Rami-Porta R, Postmus PE, Rusch V, Sobin L; International Association for the Study of Lung Cancer International Staging Committee; Participating Institutions. The IASLC Lung Cancer Staging Project: proposals for the revision of the TNM stage groupings in the forthcoming (seventh) edition of the TNM Classification of malignant tumours. J Thorac Oncol. 2007 Aug;2(8):706-14. doi: 10.1097/JTO.0b013e31812f3c1a. PMID 17762336